CLINICAL TRIAL: NCT04969822
Title: Will Embryo Selection Through Use of Artificial Intelligence (iDA) Perform Equally Compared to Day 5 Morphology?
Brief Title: eValuating iDA Selection Ability. The VISA Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitrolife (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1571 - VISA
Record Dates: First submitted 2021-06-30; First posted 2021-07-21 (Actual); Results first posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: IVF; Infertility
Keywords: Embryo; Embryo scoring; Blastocyst selection; Pregnancy rate; Live birth rate
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Embryo selection by standard morphologic criteria (No Intervention): The embryo for transfer will be selected by the embryologist on the basis of the morphologic appearances on day 5, according to the Gardner criteria using the ranking guideline.
- Embryo selection by iDA (Experimental): Time-lapse videos will be analyzed by iDA and the embryo for fresh transfer on day 5 will be prioritized on the strict basis of the embryo with the highest iDA score. For a frozen cycle; the first embryo to be warmed will be the one with the highest iDA score.
  Interventions: Device: iDAScore®

INTERVENTIONS:
Device: iDAScore® — A system that studies time lapse images obtained from the embryo culture system, Embryoscope, throughout the development to blastocyst. The system uses data acquired from a sequence of embryo images and has taught itself to identify the embryos with the highest likelihood of implanting and leading to fetal heart-beat detection.
  Arms: Embryo selection by iDA

SUMMARY:
A non-inferiority, prospective parallel group, multi-center, randomized controlled trial to investigate whether selection of a single blastocyst for transfer using the deep learning tool, iDA, results in non-inferior clinical pregnancy rate compared to trained embryologists using standard morphology criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Women undergoing IVF or ICSI with controlled ovarian stimulation with gonadotrophins and the intention to treat by either transfer of a single fresh embryo on day 5 or in case of a freeze all cycle, the first rewarmed embryo.
2. Age: Up to and including the 42nd completed birthday on the day of randomization.
3. Has at least two early blastocysts on day 5.

Exclusion Criteria:

1. Treatment involving donated eggs
2. Intention to perform any form of preimplantation genetic testing
3. The use of IMSI or polarized light in the ICSI process
4. The use of assisted hatching prior to randomization
5. Previous participation in this RCT
6. Where the cycle is carried out for fertility preservation
7. If a day 2-4 transfer is planned
8. Has a reduced likelihood of obtaining two early blastocysts on day 5 as evidenced by either: an AMH level of <3pmol/L or AFC <5 (if available)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1066 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Illingworth, A/Prof, Principal Investigator — Virtus Health, Sydney, Australia
Locations (14):
- Australia (5):
  - IVFAustralia Greenwich, Sydney, Greenwich
  - IVFAustralia Alexandria, Alexandria, New South Wales
  - IVFAustralia, Westmead, Sydney, New South Wales
  - Queensland Fertility Group (QFG), Benowa, Queensland
  - Melbourne IVF, East Melbourne, Victoria
- Denmark (3):
  - Universitetshospitalet, Aalborg
  - Aagaard Fertilitetsklinik, Aarhus
  - Regionshospitalet, Horsens
- Sweden (2):
  - Livio Gothenburg, Gothenburg
  - Reproductive medicine, Sahlgrenska University Hospital, Gothenburg
- United Kingdom (4):
  - Thames Valley Fertility (TFP), Maidenhead
  - Nurture Fertility (TFP), Nottingham
  - Oxford Fertility (TFP), Oxford
  - Wessex Fertility (TFP), Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Illingworth PJ, Venetis C, Gardner DK, Nelson SM, Berntsen J, Larman MG, Agresta F, Ahitan S, Ahlstrom A, Cattrall F, Cooke S, Demmers K, Gabrielsen A, Hindkjaer J, Kelley RL, Knight C, Lee L, Lahoud R, Mangat M, Park H, Price A, Trew G, Troest B, Vincent A, Wennerstrom S, Zujovic L, Hardarson T. Deep learning versus manual morphology-based embryo selection in IVF: a randomized, double-blind noninferiority trial. Nat Med. 2024 Nov;30(11):3114-3120. doi: 10.1038/s41591-024-03166-5. Epub 2024 Aug 9. PMID 39122964

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Embryo Selection by Standard Morphologic Criteria | Embryo Selection by iDA
Started | 533 | 533
Completed | 533 | 533
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Embryo Selection by Standard Morphologic Criteria | Embryo Selection by iDA | Total
Number analyzed (Participants) | 533 | 533 | 1066
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (3.7) | 33.8 (3.8) | 33.7 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 533 | 533 | 1066
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 41 | 37 | 78
  Denmark | 40 | 41 | 81
  United Kingdom | 106 | 112 | 218
  Australia | 346 | 343 | 689

OUTCOME MEASURES:

1. Primary Outcome: Clinical Pregnancy Rate
Description: Ultrasound evidence of an intrauterine pregnancy with a fetal heart observed
Time Frame: After 7-9 weeks of gestation
Measure: Count of Participants; unit: Participants
Arm/Group | Embryo Selection by Standard Morphologic Criteria | Embryo Selection by iDA
Number analyzed (Participants) | 533 | 533
Participants | 257 | 248

2. Secondary Outcome: Live Birth Rate
Description: Defined as the number of patients with at least one live birth after 22 completed weeks of gestation. If the exact gestational age is not known then a birth weight of ≥500gr can be used as a cut-off
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Embryo Selection by Standard Morphologic Criteria | Embryo Selection by iDA
Number analyzed (Participants) | 533 | 533
Participants | 232 | 212

3. Secondary Outcome: Positive hCG Rate Per Randomized Patient
Description: Defined as the number of patients with a positive β-hCG, determined by a hCG measurement from a blood sample or using urinary sticks
Time Frame: Tested on day 9-13 following embryo transfer
Measure: Count of Participants; unit: Participants
Arm/Group | Embryo Selection by Standard Morphologic Criteria | Embryo Selection by iDA
Number analyzed (Participants) | 533 | 533
Participants | 303 | 297

4. Secondary Outcome: Rate of Non-viable Pregnancies
Description: Defined as the difference between number of clinical pregnancies (excluding ectopic pregnancies) and number of positive β-hCG pregnancies
Time Frame: After 7-9 weeks of gestation
Measure: Count of Participants; unit: Participants
Arm/Group | Embryo Selection by Standard Morphologic Criteria | Embryo Selection by iDA
Number analyzed (Participants) | 533 | 533
Participants | 46 | 49

5. Secondary Outcome: Ongoing Pregnancy Rate
Description: Defined as the number of patients with a viable pregnancy at ≥12 weeks of gestation
Time Frame: After 7-9 weeks of gestation
Measure: Count of Participants; unit: Participants
Arm/Group | Embryo Selection by Standard Morphologic Criteria | Embryo Selection by iDA
Number analyzed (Participants) | 533 | 533
Participants | 241 | 229

ADVERSE EVENTS:
Time Frame: Adverse events were recorded up to the date of live birth, i.e. 9 months after embryo transfer.
Arm/Group | Embryo Selection by Standard Morphologic Criteria | Embryo Selection by iDA
All-Cause Mortality (participants affected / at risk) | 0/533 | 0/533
Serious Adverse Events (participants affected / at risk) | 0/533 | 0/533
Other Adverse Events (participants affected / at risk) | 0/533 | 0/533

LIMITATIONS AND CAVEATS:
The time-to-pregnancy and cumulative live birth rates were not assessed, as only the first embryo was prioritized for transfer.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT04969822/Prot_001.pdf
  • Statistical Analysis Plan (2022-11-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT04969822/SAP_000.pdf